CLINICAL TRIAL: NCT04369638
Title: Fabrication of NAM Appliance in CLP From Digital MRI Face Scan
Brief Title: Fabrication of Naso-alveolar Molding (NAM) Appliance in Cleft Lip and Palate (CLP) From Digital Magnetic Resonance Imaging (MRI) Face Scan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Brett Thomas Chiquet, Resident, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HSC-DB-20-0268
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Cleft Lip and Palate
Keywords: nasoalveloar molding; 3D printing; MRI
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 3D NAM (Experimental)
  Interventions: Device: 3D NAM; Device: Traditional NAM
- Traditional NAM (Active Comparator)
  Interventions: Device: 3D NAM; Device: Traditional NAM

INTERVENTIONS:
Device: 3D NAM — After consent and birth of the child, a face MRI will be taken of the newborn before discharge from the hospital utilizing the "feed and swaddle" technique. The MRI will be sent to the dental team to convert into a format compatible with 3D software. With the image, a NAM appliance will be digitally fabricated and 3D printed. The 3D printed model will be tested for fit on stone model made from traditional impression. Both traditional NAM and 3D printed NAM will be inserted at delivery appointment. Fit will be assessed of both appliances by applying a try-in paste to the intaglio surface and counting the number of spots needing adjustment.
Device: Traditional NAM — The patient will be seen for visit at the clinic for traditional intraoral impression and a dental stone model will be poured. An acrylic NAM will be fabricated on the stone model. The 3D printed model will be tested for fit on stone model made from traditional impression. Both traditional NAM and 3D printed NAM will be inserted at delivery appointment. Fit will be assessed of both appliances by applying a try-in paste to the intaglio surface and counting the number of spots needing adjustment.

SUMMARY:
The purpose of this study is to fabricate a nasoalveolar molding (NAM) appliance that is digitally fabricated and 3 dimensionally printed utilizing an MRI face scan and to assess the fit of the NAM in new borns with cleft lip and palate.

ELIGIBILITY:
Inclusion Criteria:

* new born babies with cleft lip and/or palate
* will undergo treatment with UT Pediatric Dental Clinic with a NAM appliance

Exclusion Criteria:

* Patients without cleft lip and/or palate
* patients that cannot tolerate an intraoral appliance
* patients that are not able to be discharged from the hospital 2-3 days after birth.

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Fit as measured by number of adjustments to the device | One month after MRI

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Wehr, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No